CLINICAL TRIAL: NCT03493815
Title: A Randomized Controlled Trial of Ultrasound-Guided Intrauterine Device (IUD) Insertion
Brief Title: A RCT of Ultrasound Guided IUD Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Stephanie Estes, Assistant Professor, Director, Robotic Surgical Services, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00008432
Record Dates: First submitted 2018-03-26; First posted 2018-04-11 (Actual); Results first posted 2020-05-11 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: IUD Not Visible

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transabdominal Ultrasound Guided IUD Insertion (Experimental): Ultrasound Guided IUD Insertion: Comparing the utility of ultrasound-guided intrauterine device (IUD) insertion compared to traditional blind insertion
  Interventions: Procedure: Transabdominal Ultrasound Guided IUD Insertion
- Traditional Blind IUD Insertion (Active Comparator): Traditional blind IUD insertion: Comparing the utility of ultrasound-guided intrauterine device (IUD) insertion compared to traditional blind insertion
  Interventions: Procedure: Traditional Blind IUD Insertion

INTERVENTIONS:
Procedure: Transabdominal Ultrasound Guided IUD Insertion — Comparing the utility of ultrasound-guided intrauterine device (IUD) insertion compared to traditional blind insertion
  Arms: Transabdominal Ultrasound Guided IUD Insertion
Procedure: Traditional Blind IUD Insertion — Comparing the utility of ultrasound-guided intrauterine device (IUD) insertion compared to traditional blind insertion
  Arms: Traditional Blind IUD Insertion

SUMMARY:
To determine the utility of ultrasound guided IUD insertion compared to the traditional blind insertion at an academic health institute where the skill level of the provider can vary greatly. We hypothesize that ultrasound-guided insertion will lead lower IUD discontinuation rates and greater patient satisfaction.

DETAILED DESCRIPTION:
(Visit 1) All interested women undergoing a scheduled IUD insertion will be screened for inclusion/exclusion criteria by the study coordinator or investigator prior to their clinic visit.

(Visit 2) After meeting eligibility criteria and being consented for the study, a subject will be ready to be randomized. Subject in both groups will fill out a visual analogue score (VAS) before and after the procedure grading their pain. Subjects will be instructed to call the investigator if they experience any abnormal uterine bleeding or problems with their IUD.

Subjects will then be randomized to one of two groups:

Group A: traditional blind IUD insertion. Group B: transabdominal ultrasound guided IUD insertion. Subjects will be randomized to either US guided or traditional placement of IUD using 1:1 allocation. The randomization scheme for this study will use variable-size, random permuted blocks where the variable block sizes are 2,4 and 6.

(Visit 3) Subjects will be scheduled to return to REI clinic 4-6 weeks (Visit 2) after insertion of the IUD as routine follow-up. Subjects will be asked about any adverse events. A routine string check in the form of a speculum exam will be performed in addition to a transvaginal ultrasound to confirm positioning of the IUD. If malposition is determined, then routine care will be to remove the IUD. The ultrasound operator will be blinded to the subject's arm in the study

(Visit 4) At 6 months subjects will be scheduled to return to REI clinic to have an IUD string check and if no strings are visualized then this will be categorized as malposition and the investigator will continue with routine care and work up Subjects who return to clinic for Visit 4 will also have a transvaginal ultrasound performed.

If the subject does not present for a clinic follow up, then she will be contacted by the Study Coordinator or investigator via phone to see if they still have their IUD in place (and when it was removed or lost).

All subjects will be surveyed for pain with the VAS and any adverse events (including abnormal uterine bleeding) will be recorded. All subjects will be asked to categorically rate their satisfaction with the IUD on a Likert Scale.

The total duration of the study is 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing IUD Insertion in an Office Setting
* Fluent in Spoken and Written English
* Premenopausal

Exclusion Criteria:

* Less than 6 Weeks Postpartum at Time of IUD Insertion
* Intraoperative IUD Insertion
* Pregnant
* Prisoners
* Cognitive Impairment
* Unable to Read or Write

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Estes, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transabdominal Ultrasound Guided IUD Insertion | Traditional Blind IUD Insertion
Started | 42 | 43
Completed | 33 | 32
Not Completed | 9 | 11

BASELINE CHARACTERISTICS:
Population: Four subjects (2 per group) were randomized but unable to insert IUD and therefore were excluded from analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Transabdominal Ultrasound Guided IUD Insertion | Traditional Blind IUD Insertion | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (6.2) | 31.5 (7.7) | 31.1 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 41 | 81
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 35 | 35 | 70
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White vs. non-white: White | 35 | 35 | 70
  White vs. non-white: Non-white | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had IUD Removed Within 6 Months
Description: IUD discontinuation rates during the 6-month post-insertion period
Time Frame: 6 Months
Population: Participants who had an IUD inserted and either discontinued the IUD or continued the IUD until the 6m visit were included. Participants who were lost to followup (outcome unknown) were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Transabdominal Ultrasound Guided IUD Insertion | Traditional Blind IUD Insertion
Number analyzed (Participants) | 33 | 32
Participants | 6 | 8
Statistical Analysis 1: Comparison: Transabdominal Ultrasound Guided IUD Insertion vs Traditional Blind IUD Insertion; Test type: Superiority; p = 0.51, binary regression w/ comp log-log link; Risk Ratio (RR) = 0.73, 95% CI 2-sided [0.28 to 1.90] — Ultrasound guided is the numerator and traditional is the denominator

2. Secondary Outcome: Number of Participants With Malpositioned IUD at 4-6 Week Visit
Description: String check in the form of a speculum exam in addition to a transvaginal ultrasound to confirm positioning of the IUD
Time Frame: 4-6 Weeks Post Insertion String Check
Population: This analysis includes participants active in the study at the 4-6 week visit. Study participants who discontinued their IUD prior to this visit, or who were lost to followup prior to this visit, were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Transabdominal Ultrasound Guided IUD Insertion | Traditional Blind IUD Insertion
Number analyzed (Participants) | 32 | 37
Participants | 3 | 6
Statistical Analysis 1: Comparison: Transabdominal Ultrasound Guided IUD Insertion vs Traditional Blind IUD Insertion; Test type: Superiority; p = 0.41, binary regression w/ comp log-log link; Risk Ratio (RR) = 0.58, 95% CI 2-sided [0.15 to 2.18] — Ultrasound guided is the numerator and traditional is the denominator

3. Secondary Outcome: Change in Pain Score
Description: Pain was assessed pre and post-insertion with a visual analog scale (VAS) ranging from 0-10 with 0 being no pain and 10 being the worst. Change in pain score was calculated as post minus pre, hence the higher the number, the greater increase in pain.
Time Frame: pre and post-insertion (both collected during the insertion visit)
Population: All participants for whom IUD was inserted.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transabdominal Ultrasound Guided IUD Insertion | Traditional Blind IUD Insertion
Number analyzed (Participants) | 40 | 41
units on a scale | 2.3 (2.5) | 2.1 (2.0)
Statistical Analysis 1: Comparison: Transabdominal Ultrasound Guided IUD Insertion vs Traditional Blind IUD Insertion; Test type: Superiority; p = 0.76, t-test, 2 sided

4. Secondary Outcome: Number of Participants Satisfied With IUD at 6 Months
Description: Satisfaction with IUD was initially assessed using a 5-point likert scale where 1=not at all happy and 5=very happy. The likert scale was then collapsed to a binary outcome of satisfied (likert scale scores 4 and 5) vs. not satisfied (likert scale scores 1,2,3).
Time Frame: 6 Months
Population: Participants who completed the 6m followup visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Transabdominal Ultrasound Guided IUD Insertion | Traditional Blind IUD Insertion
Number analyzed (Participants) | 27 | 25
Participants | 24 | 21
Statistical Analysis 1: Comparison: Transabdominal Ultrasound Guided IUD Insertion vs Traditional Blind IUD Insertion; Test type: Superiority; p = 0.70, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 6-month post-insertion period.
Description: Investigators assessed for adverse events at each visit.
Arm/Group | Transabdominal Ultrasound Guided IUD Insertion | Traditional Blind IUD Insertion
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/41
Serious Adverse Events (participants affected / at risk) | 1/40 | 0/41
Other Adverse Events (participants affected / at risk) | 19/40 | 20/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transabdominal Ultrasound Guided IUD Insertion (N=40) | Traditional Blind IUD Insertion (N=41)
malpositioned IUD (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Malpositioned IUD resulting in hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transabdominal Ultrasound Guided IUD Insertion (N=40) | Traditional Blind IUD Insertion (N=41)
Vaginal bleeding (Reproductive system and breast disorders) | 15 (16) | 16 (16)
Pelvic Pain (Reproductive system and breast disorders) | 5 (5) | 8 (8)
Heavy or prolonged menses (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Hormonal side effects (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bloating (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/15/NCT03493815/Prot_SAP_ICF_000.pdf